CLINICAL TRIAL: NCT04303832
Title: Exercise Interventions of Eye Muscles Post Strabismus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amany Refaat Mohamed Abdel Wahid, assistant lecturer, Cairo University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/001903
Record Dates: First submitted 2020-03-04; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Strabismus; Amblyopia
Keywords: Strabismus and amplyobia and physiotherapy eye exercise
MeSH Terms: conditions — Strabismus; Amblyopia | interventions — Eyeglasses

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eye exercise group (Experimental): This group made different types of eye exercises beside the traditional treatment of strabismus which is eye glasses
  Interventions: Other: eye exercises; Device: eye glasses
- control group (Sham Comparator): This group had traditional treatment of strabismus which is eye glasses
  Interventions: Device: eye glasses

INTERVENTIONS:
Other: eye exercises — Eye exercises for correcting eye deviation
  Arms: eye exercise group
Device: eye glasses — Eye glasses for correcting eye deviation

SUMMARY:
It will be hypothesized that:

* Eye exercises have a positive effect on correction of remaining ocular deviation post strabismus surgery.
* Eye exercises have a positive effect on improving amplyobia.

DETAILED DESCRIPTION:
This study applied to determine the effect of physiotherapy exercises on correction the remaining ocular deviation which still present following the strabismus surgery and also its effect on amplyobia.

Different type of physiotherapy exercises was applied to experimental group for 12 weeks beside the medical treatment applied post-surgery while the control group received traditional treatment only.

The near and far angles of ocular deviation were measured before and after the treatment for evaluation of strabismus and measuring visual acuity for evaluation of amplyobia.

ELIGIBILITY:
Inclusion Criteria:

* Patients received strabismus operation
* All types of strabismus surgery will be included
* They selected from Outpatient Clinic
* Patients begin the training program after 2 weeks of operation or more than this
* The patient still suffering from amblyopia post strabismus surgery

Exclusion Criteria:

* Muscular disorders that will impair performance during training.
* Neurological disorders.
* Malignant conditions.
* Psychiatric illness, severe behavior or cognitive disorders. Children who can't understand the therapist's instructions and orders.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
change in angle of deviation | pre and post 12 weeks
  deviation of the eye in direction rather than its normal position

SECONDARY OUTCOMES:
change in visual acuity | pre and post 12 weeks
  measure the ability of the eye to see the objects

CONTACTS AND LOCATIONS:
Overall Officials: Amany Abdel Wahid, M.Sc, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
information about statistical analysis and study report will be sheared with other researcher later on
Supporting Information: SAP, CSR
Time Frame: later on
Access Criteria: for physical therapist and ophthalmologist